CLINICAL TRIAL: NCT06780254
Title: A Two-Part Randomized Double-Blinded Placebo-Controlled, Phase 1 Study of Single and Multiple Ascending Doses of MH-001 in Healthy Participants
Brief Title: A Study to Evaluate the Pharmacokinetics (PK), Safety and Tolerability of Single- and Multiple-Ascending Doses of MH-001 in Healthy Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vespina Lifesciences Inc. (Industry)
Collaborators: Syneos Health (Other); PrimeVigilance Ltd., UK (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: MH001-01
Record Dates: First submitted 2025-01-07; First posted 2025-01-17 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: Healthy Volunteers; First In Human; Safety; Tolerability; Pharmacokinetics; Pharmacodynamics

STUDY DESIGN:
Intervention Model Description: SAD: Single Ascending Dose, 5 cohorts of different dosages versus placebo MAD: Multiple Ascending Dose, 3 cohorts of different dosages versus placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MH-001 (Experimental): In each cohort, 6/8 participants will be exposed to 1 or multiple administrations of a specific dosage of MH-001
  Interventions: Drug: MH-001
- Placebo (Placebo Comparator): In each cohort, 2/8 participants will be exposed to 1 or multiple administrations of a placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MH-001 — capsules
  Arms: MH-001
Drug: Placebo — capsules
  Arms: Placebo

SUMMARY:
First-in-Human study to demonstrate the safety and tolerability of single- and multiple-ascending doses of MH-001 in Healthy Volunteers (HVs)

ELIGIBILITY:
Inclusion Criteria:

* Male or non-childbearing potential Female, non smoker, with a Body Mass Index (BMI) between 18.5 and 32.0 kilogram per meter square (kg/m2) and red blood cells greater or equal (≥) to 120 grams per liter (g/L) for women and ≥135 g/L for men
* In good health, determined by no clinically significant findings of skin, dental, neurological, endocrine, cardiovascular, respiratory, hematological, immunological, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease

Exclusion Criteria:

* Have a history or presence of clinically significant medical illness including, but not limited to, any cardiovascular, hepatic, respiratory, hematological, chronic or relevant acute infections, relevant immunodeficiency, renal, endocrine, psychiatric or neurological disease, or any clinically significant laboratory abnormality that, in the judgment of the Investigator, indicates a medical problem that would preclude study participation.
* History of skin disorders including clinically significant active skin disease.
* History/signs and symptoms of current or recurrent teeth and gums disease
* Clinically significant abnormal laboratory test results or positive hepatitis panel and/or positive human immunodeficiency virus test.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2025-03-21 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with treatment-emergent adverse events (TEAEs) | SAD: From day of dosing until 15 days after drug administration; MAD: From first day of dosing up to 28 days after the last day (Day 28) of study drug administration
  Percentage of participants with treatment-emergent adverse events (TEAEs)

SECONDARY OUTCOMES:
Area under the concentration-time curve (AUC) of the analyte in plasma over time | SAD: Pre-dose and at multiple timepoints post-dose on Days 1 to 15; MAD: Pre-dose and at multiple timepoints post-dose on Days 1 to 56
Peak Plasma Concentration (Cmax) of the analyte in plasma | SAD: Pre-dose and at multiple timepoints post-dose on Days 1 to 15; MAD: Pre-dose and at multiple timepoints post-dose on Days 1 to 56
Time to reach Peak Concentration (Tmax) of the analyte in plasma | SAD: Pre-dose and at multiple timepoints post-dose on Days 1 to 15; MAD: Pre-dose and at multiple timepoints post-dose on Days 1 to 56

CONTACTS AND LOCATIONS:
Locations (1):
- Syneos Health clinic, Québec, Quebec, Canada